CLINICAL TRIAL: NCT06161311
Title: The Influence of Baseline Relative Peripheral Refraction in Myopia Control Using Myopic Defocus
Brief Title: Baseline Relative Peripheral Refraction in Myopia Control
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Centre for Eye and Vision Research (Other); HOYA Lamphun Ltd (Industry)
Responsible Party: Principal Investigator, LEUNG Tsz Wing, Research Assistant Professor, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HSEARS20221229003-01
Record Dates: First submitted 2023-11-30; First posted 2023-12-07 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2023-11

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Myopic RPR group (Active Comparator): Patients with myopic relative peripheral refraction
  Interventions: Device: DIMS lenses
- Hyperopic RPR group (Active Comparator): Patients with hyperopic relative peripheral refraction
  Interventions: Device: DIMS lenses

INTERVENTIONS:
Device: DIMS lenses — Defocus incorporated multiple segments lenses, which use induce peripheral myopic defocus to control for myopia development in children

SUMMARY:
Myopia has become a world concern and its prevalence has increased in recent decades. Myopic defocus has been applied for slowing down the axial elongation and myopia progression, which is mainly based on the theory of simultaneous competing defocus and peripheral optics. Defocus Incorporated Multiple Segments (DIMS) spectacle lenses impose myopic defocus in the central or peripheral retina, with myopia progression being retarded by 50% to 60%. However, the optimal amount of myopic defocus has not yet been determined. Relative peripheral refraction (RPR) is used to indicate the difference between peripheral refraction and central refraction. Previous studies showed that retinal shape determined RPR, and baseline RPR may influence the myopia control efficacy using DIMS lenses on myopic children. It is still unclear if any other unknown factor influenced the final myopia control outcome in these young children with myopic RPR at baseline. Unlike our previous study8 that bias on hyperopic RPR children (myopic RPR, n = 27; hyperopic RPR, n = 52), this study is a case-control study with the same sample size for each RPR group. We will also include younger children who are more prone to have myopic RPR and develop high myopia. The results should provide new insight into the myopia control strategy in early-onset myopic children.

In the current study, we will investigate the influence of baseline RPR in myopia retardation using DIMS lenses among young myopic children.

This will ba a 1-year prospective clinical trial. Through G*Power (version 3.1.9.6) calculation, 80 healthy myopic subjects (40 myopic RPR vs 40 hyperopic RPR) aged 5-9 years should be needed. After screened by inclusion criteria, eligible participants will be assigned to wear DIMS lenses for 1 year (12 months, 8 hour per day, 7 days per week). This study includes 5 visits: Visit 1: baseline, Visit 2: lens dispensing, Visit 3: 2-week follow-up, Visit 4: 6-month follow-up, and Visit 5: 12-month follow-up. All eye examinations will be carried out in the Optometry Research Centre (A137), the School of Optometry, the Hong Kong Polytechnic University. The main data collection, including refractive error, axial length, related ocular parameters will be measured at baseline, 6-month and 1-year visits. At the lens dispensing and 2-week follow-up visits, vision acuity testing and computer scanning of posterior eyes will be measured. New DIMS lens will be replaced and upgraded if the equivalent sphere of refraction (SER) is changed or visual acuity change.

The following data will be statistically analyzed. The primary outcome data include the difference in change in SER with cycloplegia between the myopic and hyperopic RPR from the baseline over 12 months of treatment. Secondary outcomes data include the changes in axial length, peripheral refraction, relative peripheral refraction, the amplitude of accommodation, lag of accommodation, corneal curvature, phoria and stereoacuity.

ELIGIBILITY:
Inclusion Criteria:

* Age at enrolment: 6-9 years
* Spherical equivalent refraction (SER): -0.75 to -5.00 Diopters (D)
* Astigmatism: -1.50 D or less
* Anisometropia: 1.50 D or less
* Spectacle best-corrected monocular visual acuity (VA): 0.00 logMAR or better

Exclusion Criteria:

* Ocular and systemic abnormalities might affect visual functions or refractive development
* Prior use of any drugs or optical devices of myopia control treatment.

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-04-03 (Estimated); Study Completion 2025-04-03 (Estimated)

PRIMARY OUTCOMES:
Cycloplegic refractive error | Baseline; 2 weeks, 6 months and 12 months post-treatment
  Refractive error measured after instillation of cycloplegia

SECONDARY OUTCOMES:
Axial length | Baseline; 2 weeks, 6 months and 12 months post-treatment
  Length of the eye
Peripheral refraction | Baseline; 2 weeks, 6 months and 12 months post-treatment
  Refractive errors at peripheral fields
Amplitude and lag of accommodation | Baseline; 2 weeks, 6 months and 12 months post-treatment
  Ability of the eyes to accommodate
Corneal curvature | Baseline; 2 weeks, 6 months and 12 months post-treatment
  Power of the cornea
Phoria and stereoacuity | Baseline; 2 weeks, 6 months and 12 months post-treatment
  Coordination of the two eyes

CONTACTS AND LOCATIONS:
Locations (1):
- Optometry Research Clinic, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided